CLINICAL TRIAL: NCT00318305
Title: Patient Preference and Acceptance With Sodium Phosphate Tablet Preparation for Colonoscopy: A Prospective Study
Brief Title: Patient Preference With Visicol Tablet Preparation for Colonoscopy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: InKine Pharmaceutical (Industry)
Responsible Party: Suryakanth Gurudu, MD, Mayo Clinic
Other Study IDs: 392-05
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Preparation for Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine patient preference and acceptance of tablet sodium phosphate bowel preparation in patients who had polyethylene glycol (PEG) solution for their prior colonoscopy. This study will provide answers related to the patient preferences and their acceptance of this new method of bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* Prior colonoscopy with PEG solution in the past one year
* Must be able to swallow tablets

Exclusion Criteria:

* Patients below 18 years and above 100 years.
* Congestive heart failure
* Chronic renal failure
* Pre-existing electrolyte disorder
* Pre-existing mega-colon or a motility disorder.
* Patients with pre-existing seizure disorder.
* Patients scheduled for colonoscopy after 1:00 p.m. will be excluded from the study.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Scheduled colonoscopy list will be reviewed to identify potential subjects for recruitment. A cover letter will be sent to the potential study subject with tablet preparation as an alternative to Golytely preparation ( PEG). For subjects who are willing to participate, a prescription for 28 tablet sodium phosphate bowel preparation as outlined in appendix: A will be mailed. A questionnaire will be given to the patients prior to their colonoscopy to identify their preferences regarding bowel preparation and their acceptance ( see appendix: B).
  A separate validated questionnaire will be given to participating physicians after the procedure, to quantitate the colonic cleansing (appendix : C). Adverse events will be documented. A statistical analysis of the results will be done at the end of the study.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2005-03; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suryakanth R. Gurudu, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States